CLINICAL TRIAL: NCT05083221
Title: The Effectiveness of an Aural Rehabilitation Program on Communication Abilities, Depression, Loneliness and Quality of Life in Older Adults With Hearing Impairment
Brief Title: Effect of an Aural Rehabilitation Program in Hearing-impaired Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202007027RINA
Record Dates: First submitted 2021-09-13; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Older Adults; Hearing Impairment; Nursing
Keywords: audiological rehabilitation; hearing impairment; quality of life; older adults; communication ability; depression; loneliness
MeSH Terms: conditions — Hearing Loss; Depression

STUDY DESIGN:
Intervention Model Description: In this single-blind, randomized controlled trial, older adults aged 65 years or older with hearing impairment will be randomized into either the intervention group (Hear-Talk-Activity intervention group) or the control group (waitlist control group)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hear-Talk-Activity audiological rehabilitation program (Experimental): Audiological intervention program
  Interventions: Behavioral: Hear-Talk-Activity audiological program
- Control group (No Intervention): Waitlist control program

INTERVENTIONS:
Behavioral: Hear-Talk-Activity audiological program — The participants were randomly assigned to either the experimental group or the waiting-list control group, using a computer-generated list of random numbers.
  Arms: Hear-Talk-Activity audiological rehabilitation program

SUMMARY:
Hearing impairment in older adults is becoming a common health problem as the population ages. The impact of hearing impairment in older adults includes not only physical function and cognitive performance, but also depression, loneliness and social isolation, as well as having a negative impact on quality of life and financial status. Therefore, an audiological rehabilitation program intervention is recommended. The purposes of this study are to examine the effects of an audiological rehabilitation program (Hear-Talk-Activity audiological rehabilitation program) intervention on communication abilities, depression, loneliness and quality of life outcomes in older adults with hearing impairment. The single-blind, randomized control trial will include older adults aged 65 years or older with hearing impairment and aid user. Participants will be randomized to either intervention groups or control groups.

DETAILED DESCRIPTION:
The study will be an experimental design featuring repeated measures, with data collected from a pretest, a posttest and a follow-up test. An estimated total of 96 participants will be randomly assigned to experimental and control groups. The experimental group will participate in a 10-week aural rehabilitation program (Hear-Talk-Activity audiological rehabilitation program), including provide information, hearing aids and assistive listening devices, communication strategies and skills, personal coping and adjustment, psychosocial support and stress management, consisting of 60-minute sessions once per week, while the control group will be put on a waiting-list group. Each group will be assessed of the outcomes at 3 time points: baseline (T0), three months following the intervention (T1) and again at six months following the intervention (T2). The investigators will use the Hearing Handicap Inventory for the Elderly-Screening version (HHIE-S), the 10-item version of the Center for Epidemiological Studies Depression Scale (10-item CES-D), the short-form University of California, Los Angeles (UCLA) Loneliness Scale-8 item (ULS-8) and the Short Form-12 health survey (SF-12) as the outcome indicators. The principle of intention-to-treat (ITT) analysis will be used, and the result will be analyzed mainly by generalized estimating equation (GEE).

ELIGIBILITY:
Inclusion Criteria:

* being 65 or older
* Pure-Tone Average (PTA) more than 40 decibel (dB) Hearing Level (HL) and aid users less than half a year
* living in the community
* having normal cognitive
* articulate in the Mandarin Chinese language
* signing a consent form to participate

Exclusion Criteria:

* severe psychiatric disorders
* acoustic neuroma lead to hearing impairment
* chronic otitis media lead to hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline the Hearing Handicap Inventory for the Elderly-Screening version at 3 months, and 6 months | baseline, 3th, 6th month
  A score of participants in baseline communication abilities as assessed by the Hearing Handicap Inventory for the Elderly-Screening version. The overall score ranging from 0 to 40, which higher scores indicating poorer communication abilities
Change from Baseline the 10-item version of the Center for Epidemiological Studies Depression Scale at 3 months, and 6 months | baseline, 3th, 6th month
  A score of participants in baseline depression as assessed by the 10-item version of the Center for Epidemiological Studies Depression Scale. The overall score ranging from 0 to 30, which higher scores indicating severe depression
Change from Baseline the short-form UCLA Loneliness Scale-8 item at 3 months, and 6 months | baseline, 3th, 6th month
  A score of participants in baseline loneliness as assessed by the short-form UCLA Loneliness Scale-8 item. The overall score ranging from 8 to 32, which higher scores indicating severe loneliness
Change from Baseline the Short Form-12 health survey at 3 months, and 6 months | baseline, 3th, 6th month
  A score of participants in baseline quality of life as assessed by the Short Form-12 health survey. The overall score ranging from 0 to 100, which higher scores indicating better quality of life
Change from Baseline the International Outcome Inventory for Hearing Aids at 3 months, and 6 months | baseline, 3th, 6th month
  A score of participants in baseline communication abilities and aids satisfaction as assessed by the International Outcome Inventory for Hearing Aids. The overall score ranging from 7 to 35, which higher scores indicating better communication abilities and aid satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Meei-Fang Lou, Ph.D., Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng YC, Chang NT, Liu SH, Gau BS, Liu TC, Lou MF. Effects on health outcomes following a nurse-led hearing loss management intervention designed for older adults: A randomized controlled trial. Int J Nurs Stud. 2025 Jun;166:105050. doi: 10.1016/j.ijnurstu.2025.105050. Epub 2025 Mar 11. PMID 40157018